CLINICAL TRIAL: NCT00809094
Title: A Multi-Center, Phase IIB, Randomized, Placebo-controlled, Double-Blind Study Of The Effects Of N-Acetylcysteine On Redox Changes and Lung Inflammation In Cystic Fibrosis Patients
Brief Title: NAC Phase IIB: A Multi-Center, Phase IIB, Randomized, Placebo-controlled, Double-Blind Study Of The Effects Of N-Acetylcysteine On Redox Changes and Lung Inflammation In Cystic Fibrosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-12112008-1378
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo was administered oral tablet TID for 24 weeks.
  Interventions: Drug: Placebo
- N-Acetylcysteine (Active Comparator): Participants received 900 mg of oral N-acetylcysteine TID for 24 weeks.
  Interventions: Drug: N-acetylcysteine (NAC)

INTERVENTIONS:
Drug: N-acetylcysteine (NAC)
  Other Names: PharmaNAC
  Arms: N-Acetylcysteine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This Phase IIB proof-of-concept study would examine the effects of an investigational product called N-acetylcysteine (NAC) on the basic processes that cause inflammation in CF lung disease. We hope to learn more about the causes of lung disease in cystic fibrosis by studying the characteristics of the inflammation in the lungs of patients who have CF.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 7 years of age or older
2. Diagnosis of CF based upon the following criteria:

   1. One or more clinical features characteristic of CF AND (b or c)
   2. Positive sweat test > 60 mEq/L by quantitative pilocarpine iontophoresis
   3. A genotype with two identifiable mutations consistent with CF
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative
4. Clinically stable with no evidence of acute upper or lower respiratory tract infection within 4 weeks prior to enrollment
5. Stable mild or moderately severe lung disease defined by an FEV1 > or = 40% and < or = 85% predicted for age based on the Wang (males < 18 years, females < 16 years) or Hankinson (males > or = 18 years, females > or = 16 years) standardized equations
6. Able to tolerate sputum induction with 3% hypertonic saline and to expectorate
7. Able to perform repeatable, consistent efforts in pulmonary function testing
8. Weight > or = 25 kg at time of enrollment
9. Females of child bearing potential must be willing to use birth control (IUD, oral, transdermal, or parenteral contraceptives; abstinence)

Exclusion Criteria:

1. Clinically significant liver enzymes (AST, ALT or GGT) > 2.5 times the upper limit of normal at screening
2. History of ABPA, unless have evidence of a stable IgE (< 5% increase compared to previous test) for 6 months prior to enrollment
3. Current or history of rheumatic or collagen vascular disorders
4. Use of NSAIDS other than for chronic therapy within 1 week prior to enrollment
5. Initiation of chronic therapy with ibuprofen, azithromycin, TOBI® or Aztreonam within 6 weeks prior to enrollment
6. Consumption or inhalation of antioxidants (including NAC, GSH, Immunocal, Nacystelyn, pentoxyfilline) within 6 weeks prior to enrollment
7. Use of oral or IV corticosteroids within 4 weeks prior to enrollment
8. Use of acetaminophen within 3 days prior to enrollment
9. Unable to forego during the study:

   * Vitamin E: more than 400 IU/day for subjects < or = 12 years of age and 800 IU/day for subjects > 12 years of age
   * Vitamin C: more than 0.5 gm/day
   * More than two alcoholic drinks per day
10. Known hypersensitivity to oral PharmaNAC®
11. Current cigarette consumption
12. Pregnant or breastfeeding
13. Subject unlikely to complete the study as determined by the Investigator
14. Any condition that the Investigator believes would interfere with the intent of this study or would make participation not in the best interest of the subject
15. Participation in trials for other anti-inflammatory or therapeutic investigational drugs within 6 weeks prior to enrollment

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol K. Conrad, Principal Investigator — Stanford University
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University School of Medicine, Stanford, California
  - National Jewish Hospital, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Shands at the University of Florida, Gainesville, Florida
  - Columbia University Medical Ctr, New York, New York
  - Duke Children, Durham, North Carolina
  - The PennState Milton S Hersey Medical Ctr, Hershey, Pennsylvania
  - The Children, Philadelphia, Pennsylvania
  - Children, Pittsburgh, Pennsylvania
  - University of Utah, Primary Children, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 11/4/2008. Recruitment process was staggered: Stanford cohort first to focus on safety data related to potential pulmonary hypertension. After half of the Stanford cohort reached the 8-week time point, the DSMC evaluated PH safety data. The other sites then began enrollment. Final subject enrolled on 2/2011.
Groups:
- Study Drug: N-acetylcysteine (NAC) :PharmaNAC® 900 mg effervescent tablets in blister packs were supplied by BioAdvantex Pharma, Inc. (Mississauga, ON, Canada).
- Placebo: Identically packaged effervescent tablets that contained only the carrier were provided in blister packs by BioAdvantex Pharma, Inc. (Mississauga, ON, Canada)
Period: Overall Study
Arm/Group | Study Drug | Placebo
Started | 36 | 34
Completed | 36 | 33
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug | Placebo | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 10 | 19
  Between 18 and 65 years | 27 | 24 | 51
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in the Logarithm of the Level of Human Neutrophil Elastase (HNE) Activity Measured in Sputum
Description: (change in log10 HNE in the active treatment group) - (change in log10 HNE in the placebo group)
Time Frame: From enrollment to end of the 24-week trial
Population: The primary endpoint analyses described uses the subset of the ITT population with complete case data. 70 subjects randomized, 65 completed the Week 12 visit and 62 completed the study. There were 6 withdrawals in the NAC group and 2 in Placebo. Five out of 6 subjects in the NAC group withdrew due to subject decision. Missing data was not imputed.
Measure: Log Mean (95% Confidence Interval); unit: log10 mcg/mL
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 26 | 30
log10 mcg/mL | 0.03 [-1.12 to 1.38] | -0.17 [-1.20 to 0.67]
Statistical Analysis 1: Comparison: Study Drug vs Placebo; Null hypothesis: there will be no difference in the change in human neutrophil activity measured from baseline to end of the study (24 weeks); Test type: Superiority or Other; p = 0.14, t-test, 2 sided; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.07 to 0.48]

2. Secondary Outcome: Change in FEV1 (Percent of Predicted for Age)
Description: Change in forced expiratory volume in 1 second as compared to normals for age (percent of predicted)
Time Frame: From enrollment to the end of the 24-week trial
Population: Out of 70 subjects randomized, 65 completed the Week 12 visit and 62 completed the study. There were 6 withdrawals in the NAC group and 2 in Placebo. Five out of 6 subjects in the NAC group withdrew due to subject decision. Missing data was not imputed.
Measure: Number (95% Confidence Interval); unit: percent of predicted vlaues
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 30 | 32
percent of predicted vlaues | 1.055 [-26.16 to 25.73] | -5.62 [-24.54 to 19.69]

3. Secondary Outcome: FEV1 (L)
Description: Forced expiratory volume in 1 second (Liters)
Time Frame: Baseline to end of study (24 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Liter
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 30 | 32
Liter | 2.5 [-21.92 to 30.28] | -4.35 [-25.00 to 22.94]

4. Secondary Outcome: FEF 25-75% (L/Sec)
Description: Difference in mid-expiratory flow rates between 25 to 75% of the vital capacity, in L/sec measured at the beginning of the study to the end of the study.
Time Frame: Baseline to end of study (24 weeks)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: L/sec
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 30 | 32
L/sec | 0.08 [-0.39 to 0.88] | -0.13 [-1.22 to 0.39]

5. Secondary Outcome: FEF 25-75% (Percent of Predicted)
Description: Difference in the forced expiratory flow rate in mid-exhalation as a percent of predicted to standard values measured from baseline to the end of study (24 weeks).
Time Frame: Baseline to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percent of predicted
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 30 | 32
percent of predicted | 1.33 [-16.46 to 25.32] | -3.81 [-25.20 to 9.78]

6. Other Pre Specified Outcome: Change in DLCO (ml/Min/mmHg) Over Time by Treatment Group
Description: Change in the diffusing capacity of carbon monoxide across the lung measured from baseline to end of 24-week study.
Time Frame: Baseline to 24 weeks
Population: Sixteen subjects at Stanford University were enrolled as an initial safety cohort, and their data was used to evaluate the potential for NAC to cause PH in CF subjects.
Measure: Mean (Standard Deviation); unit: ml/min/mm Hg
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 8 | 8
ml/min/mm Hg | -0.32 (2.86) [lower limit -4.76] | -1.39 (3.93)

7. Other Pre Specified Outcome: Change in ECHO Tricuspid Regurgitation (mm Hg) Over Time by Treatment Group
Description: Change in measure of estimated right ventricular pressure over the 24-week study period
Time Frame: Baseline to 24 weeks
Population: Sixteen subjects at Stanford University were enrolled as an initial safety cohort, and their data was used to evaluate the potential for NAC to cause PH in CF subjects. 1 subject in NAC cohort has missing data. It was not imputed
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 7 | 8
mm Hg | 31.5 (6.02) | 31.75 (5.84)

ADVERSE EVENTS:
Arm/Group | Study Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 15/36 | 17/34
Other Adverse Events (participants affected / at risk) | 33/36 | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Drug (N=36) | Placebo (N=34)
Pulmonary Exacerbation (Respiratory, thoracic and mediastinal disorders) | 15 | 17 — These events were not considered related to study drug by the treating physician
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug (N=36) | Placebo (N=34)
Fatigue (General disorders) | 13 (17) | 8 (21)
Forced Expiratory Volume Decreased (Investigations) | 9 (11) | 9 (14)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 5 (6)
Constipation (Gastrointestinal disorders) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (4)
Chest Discomfort (General disorders) | 3 (5) | 5 (7)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 3 (5) | 2 (3)
Pyrexia (General disorders) | 4 (7) | 8 (14)
sinusitis (Infections and infestations) | 3 (3) | 1 (1)
Pulmonary function test decreased (Investigations) | 2 (3) | 3 (3)
Weight decreased (Investigations) | 5 (6) | 5 (6)
white blood cell count increased (Investigations) | 2 (2) | 1 (1) — s
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 3 (3)
Sinus headache (Nervous system disorders) | 4 (18) | 4 (6)
Anxiety (Psychiatric disorders) | 2 (4) | 0 (0)
Nephrolitiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (55) | 21 (45)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 6 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (16)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 13 (18)
Rales (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 8 (11)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (9)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (6)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No